CLINICAL TRIAL: NCT05049746
Title: Identifying Decision Making Needs for Older Adult Women With Breast Cancer Considering Neoadjuvant or Adjuvant Chemotherapy
Brief Title: Identifying Decision Making Needs for Older Adult Women With Stage I-III Breast Cancer Considering Neoadjuvant or Adjuvant Chemotherapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0055; NCI-2021-07005 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0055 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-02; First posted 2021-09-20 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Other): Participants in the intervention arm only will then be asked to look at the decision tool that includes educational materials about the diagnosis and treatment of breast cancer.
  These could be written information, graphics, videos, animations, or questionnaires.
  This decision tool will personalize the decision to you specifically and support your decision-making process
  Interventions: Other: Discussion; Other: Interview; Other: Questionnaire Administration
- Non-Intervention Arm (No Intervention): Participants undergo interviews and complete questionnaires over 1-2 hours. Patients and physicians also participate in a discussion and complete shared decision-making questionnaire over 15-30 minutes.

INTERVENTIONS:
Other: Discussion — Participate in discussion
  Other Names: Discuss
  Arms: Intervention Arm
Other: Interview — Participate in interview
  Arms: Intervention Arm
Other: Questionnaire Administration — Complete questionnaire
  Arms: Intervention Arm

SUMMARY:
This study collects information and identifies decision making needs for older adult women with stage I-III breast cancer considering neoadjuvant and adjuvant chemotherapy. Using this information, a decision support tool is then developed to provide patients and physicians with tailored information regarding the risks and benefits of chemotherapy and values clarification to support high-quality, shared decision. Subsequently, the decision support tool will be tested amongst older patients with early-stage breast cancer and health care providers navigating the decision process around chemotherapy, and further refined through an iterative process.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize and describe the informational needs and preferences in older adult women who intend on receiving neoadjuvant or adjuvant chemotherapy for stage I-III breast cancer.

Ia. Conduct semi-structured interviews with women who have completed the treatment decision process to collect informational needs and elicit decision-making needs and preferences.

Ib. Utilize validated data collection instruments to assess the shared decision-making process and health literacy needs.

II. To develop a decision support tool for use by patients and healthcare providers to guide the chemotherapy decision-making process in older women (>= 65) with early-stage breast cancer.

IIa. To conduct cognitive testing of the decision tool. IIb. To conduct a field test of the decision tool in order to demonstrate feasibility and acceptability in real-world clinical settings.

OUTLINE:

Patients undergo interviews and complete questionnaires over 1-2 hours. Patients and physicians also participate in a discussion and complete shared decision-making questionnaire over 15-30 minutes. Subsequently, a decision support tool will be developed consistent with standards for content development and evaluation from the International Patient Decision Aid Standards (IPDAS) Collaboration and implemented through an iterative process of design, development and evaluation to engage end users in its development. Once developed, field testing of the decision tool will be conducted to demonstrate feasibility and acceptability in real-world clinical setting, followed by pilot testing to evaluate the efficacy of the decision support tool.

ELIGIBILITY:
INCLUSION CRITERIA:

Patient Inclusion Criteria

* Women aged 65 years or older
* Must write and speak English
* Must have been diagnosed with Stage I-III breast cancer
* Must have made decision to either receive or not receive neoadjuvant or adjuvant chemotherapy
* Must be within 3 months of breast cancer neoadjuvant or adjuvant chemotherapy treatment decision
* Self-reported no visual or auditory deficits
* SUBAIM 2b: Women aged 65 years or older
* SUBAIM 2b: Must write and speak English
* SUBAIM 2b: Must have been diagnosed with stage I-III breast cancer
* SUBAIM 2b: Must be a candidate for chemotherapy or targeted therapy (in the setting of HER2+ breast cancer)
* SUBAIM 2b: Must be making a decision regarding chemotherapy
* SUBAIM 2b: Self-reported no visual or auditory deficits
* PHYSICIAN INCLUSION CRITERIA
* Physician for patient recruited to participate in study (physician criteria)

Exclusion Criteria:

None

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Decision making needs assessment questionnaire | through study completion, an average of 1 year
  The mean score of the shared decision making questionnaire and its standard deviation along with the median and the range will be computed for both the patient and physician study population. Score Range-(0-4) 0-Not at all confident 4-very confident

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Karuturi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org